CLINICAL TRIAL: NCT01371383
Title: The Effect of Omega-3 Polyunsaturated Fatty Acids in the Treatment and Prevention of Relapse of Bipolar Disorder.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Kuan-Pin, China Medical University Hospital, National Science and Technology Council, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DOH94F044
Record Dates: First submitted 2011-06-07; First posted 2011-06-10 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- n-3 fatty acids (Experimental): EPA 1680 mg/d + DHA 880 mg/d
  Interventions: Dietary Supplement: n-3 fatty acids
- Placebo (Placebo Comparator): Soybean oil
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: n-3 fatty acids — EPA 1680 mg/d + DHA 880 mg/d
  Arms: n-3 fatty acids
Dietary Supplement: placebo — Soybean oil
  Other Names: control
  Arms: Placebo

SUMMARY:
The whole study will be divided into two major parts: (A) A 12-week, double-blind, randomized controlled, parallel n-3 fatty acids adjunctive therapy study in 30 bipolar disorder patients with mild to moderate depression. (B) A double-blind, randomized controlled, parallel n-3 fatty acid add-on prophylactic study in 31 patients with stable bipolar disorder.

DETAILED DESCRIPTION:
Part of the study will be a 12-week parallel-group placebo-controlled double-blind randomized n-3 fatty acids add-on combination therapy trial. A total of 30 patients in the acute depression stage of bipolar disorder will be collected from outpatient clinics and randomly assigned to receive n-3 fatty acids or placebo. T-test (or Mann-Whitney U-Test) will be used to evaluate the differences in the severity of depressive and manic symptoms between the two groups across the study points. The second part of the study will be a 6-month add-on prophylactic trial with parallel-group, double-blind random allocation to n-3 fatty acids or placebo groups. A total of 31 patients with stable bipolar disorder recruited by newspaper advertisements will be recruited and randomly assigned to receive n-3 fatty acids or a placebo. Kaplan-Meier Survival analysis will be used to evaluate the differences in the recurrence rate of bipolar depression between the two groups. Also, t-test (or Mann-Whitney U-Test) will be used to evaluate the differences in the severity of depressive and manic symptoms between the two groups across the study points. The 2 separate studies will be conducted after approval from the Human Trials Committee.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV criteria for bipolar disorder.
2. Age being age 18-65.
3. Capacity and willingness to give written informed consent.
4. Routine biochemical parameters within normal range.

Exclusion Criteria:

1. Presence of any major medical illnesses.
2. Recent or past history of other DSM-IV axis I diagnoses such as psychotic disorders, organic mental disorders, substance abuse, substance dependence and anxiety disorder; acute psychotic state or strong suicidal attempts; and DSM-IV axis-II diagnoses, including borderline and antisocial personality disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-01-01; Primary Completion 2014-05-31 (Actual); Study Completion 2015-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in HRSD-21 scores | Weeks 0, 1, 2, 4, 6, 8, and 12
  Differences in depression severity based on the Hamilton Rating Scale for Depression 21 (HRSD) across the study points.
Differences in recurrence rate of bipolar depression | From 0 to 6 months
  Differences in the rate of recurrence of bipolar disorder between the patients in the n-3 group and placebo group across the study points.

SECONDARY OUTCOMES:
Changes in Young Mania Rating Scale scores | Weeks 0, 1, 2, 4, 6, 8, and 12
  Changes in Young Mania Rating Scale scores across the time points in the study

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Pin Su, MD PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Appleton KM, Voyias PD, Sallis HM, Dawson S, Ness AR, Churchill R, Perry R. Omega-3 fatty acids for depression in adults. Cochrane Database Syst Rev. 2021 Nov 24;11(11):CD004692. doi: 10.1002/14651858.CD004692.pub5. PMID 34817851